CLINICAL TRIAL: NCT01472653
Title: Skin Reaction to Cetuximab as Criteria for Treatment Selection in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck: Phase 2 Study
Brief Title: Treatment Selection According to Skin Reaction to Cetuximab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORL-01-11
Record Dates: First submitted 2011-10-23; First posted 2011-11-16 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck Cancer; Radiochemotherapy; Radioimmunotherapy; Skin rush; locoregional control; Survival; Toxicity
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Radiotherapy; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cisplatin — cisplatin 30 mg/m2/week I.V. during radiotherapy
Radiation: radiotherapy — 3-dimensional conformal radiotherapy planning and delivery, 35x2 Gy/day over 7 weeks
Drug: cetuximab — cetuximab 400 mg/m2 I.V. 1 week before the start of radiotherapy, cetuximab 250 mg2/week I.V. during radiotherapy
  Other Names: Erbitux

SUMMARY:
The therapy of patients with locally advanced head and neck cancer will be adjusted to the grade of skin rush as recorded after the first two cycles of Cetuximab and Cisplatin, i.e. either with radioimmunotherapy (radiotherapy and Cetuximab) or radiochemotherapy (radiotherapy and Cisplatin.

DETAILED DESCRIPTION:
Background: According to literature, the treatment results in irradiated patients who develop intensive skin reaction after concomitant Cetuximab administration appear improved as compared to the results of standard combination of radiotherapy and Cisplatin. In other patients, no beneficial effect of Cetuximab is expected and the therapy with Cisplatin (concomitantly with irradiation) is more effective in this group.

In this proposed single-institution non-randomized phase II study on patients with locally advanced squamous cell carcinoma of the head and neck, the therapy will be adjusted to the grade of skin rush as recorded after the first two cycles of Cetuximab and Cisplatin, i.e. either with radioimmunotherapy (radiotherapy and Cetuximab) or radiochemotherapy (radiotherapy and Cisplatin).

Methods: In the patients with inoperable tumors, induction chemotherapy (Docetaxel 75 mg/m2, Cisplatin 75 mg/m2, 5-Fluorouracil 750 mg/m2 in continuous infusion days 1-5; repeated every 21 days for 4 cycles) will be administered. In the week before the first fraction of radiotherapy, all patients will receive a loading dose of Cetuximab (400 mg/m2) and combination of Cetuximab (250 mg/m2) and Cisplatin (30 mg/m2) during the first week of irradiation. After multidisciplinary assessment of the grade of skin rush, conducted at the end of the second week of irradiation, the patients will be grouped as follows: arm A - skin rush of CTCAE v3.0 grade <2 will proceed with radiochemotherapy with Cisplatin; arm B - skin rush of CTCAE v3.0 grade >=2 will proceed with radioimmunotherapy with Cetuximab.

The planned number of patients included in the study is 120 (arm A - 50, arm B - 70) and recruitment period is 3 years. The primary objective of the study is to determine radiologically the complete response rate 12-14 weeks after therapy. The secondary objectives are locoregional control, progression-free survival and overall survival at 2 years after therapy, acute and late toxicity.

Expected results: The expected complete response rate in patients treated with radiochemotherapy and those treated with radioimmunotherapy is 50% and 75%, respectively. We also expect the difference in an absolute survival gain between the groups to be 25%.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma, histologically proven (with HPV-status determined in patients with oropharyngeal primary)
* Tumour site: oral cavity, oropharynx, hypopharynx or larynx.
* Locally and/or regionally operable and inoperable tumors (UICC TNM stages III, IVa or IVb), without distant metastases (M0-stage)
* Male or female ≥18 years of age
* Expected survival >6 months
* WHO performance status 0-2
* Laboratory parameters:

hemoglobin ≥100 g/L; leukocyte count > 3.5x109/L, absolute neutrophil count ≥ 1.5x109/L; platelet count > 100x109/L; total bilirubin < 1.25x upper normal limit; transaminases (ALT, AST) < 5x upper normal limit; creatinine clearance (ECC) ≥ 60 ml/minute;

* Presence of at least one bidimensionally measurable index lesion
* Effective contraception for both male and female subjects if risk of conception exists
* Signed written informed consent

Exclusion Criteria:

* Other previous malignancy within 5 years, with exception of a history of a previously adequately treated basal cell carcinoma of the skin or pre- invasive carcinoma of the cervix
* Chemotherapy ineligibility:

unstable cardiopulmonary, renal and liver disease likely to compromise the safe delivery of I.V. infusion (chemotherapy); haematologic diseases; clinically evident hearing impairment; pre-existing motor or sensory neurotoxicity grade ≥ 2 according to the CTCAE v3.0; previous administration of Cetuximab or Cisplatin;

* Active, uncontrolled infection
* Medical or psychological condition which in the opinion of the investigator precludes the safe administration of the planned radiotherapy or systemic therapy
* Known drug abuse or severe alcohol abuse
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
locoregional complete response rate | 12-14 weeks after therapy
  The primary objective of the study is to determine radiologically the complete response rate 12-14 weeks after therapy.

SECONDARY OUTCOMES:
feasibility (toxicity profile) of the proposed regimen | participants will be followed for the duration of treatment (an expected average of 20 weeks)
  number of patients with adverse events graded according to the National Cancer Institute CTC v3.0 (as measure of safety and tolerability)
locoregional control | at 2 years after thapy
  Locoregional control will be calculated from the first day of the therapy to the occurrence of the local and/or regional recurrence (whichever will occur first) or death from any cause other than distant metastasis.
progression-free survival | 2 years after therapy
  Progression-free will be calculated from the first day of the therapy to the appearance of local or regional recurrence, distant metastases, secondary primary cancer or death from any cause.
overall survival | 2 years after therapy
  Overall survival is defined as a time interval between the first day of therapy and death from any cause.
late toxicity including thyroid function | up to 2 years post-therapy
  number of patients with adverse events graded according to the National Cancer Institute CTC v3.0 (as measure of safety and tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Primož Strojan, Prof., Principal Investigator — Dept. of Radiation Oncology, Institute of Oncology Ljubljana, Slovenia; Branko Zakotnik, Prof., Principal Investigator — Dept. of Medical Oncology, Institute of Oncology Ljubljana, Slovenia
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia